CLINICAL TRIAL: NCT06081907
Title: A Prospective, Multi-cohort Study on Efficacy and Safety of IBI363 for Advanced Solid Tumors
Brief Title: The Efficacy and Safety of IBI363 in Solid Tumors
Acronym: Promise
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBI-363
Record Dates: First submitted 2023-10-05; First posted 2023-10-13 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- IBI363 DL1 (Experimental): IBI363 + IBI325
  Interventions: Drug: IBI363
- IBI363 DL2 (Experimental): IBI363 + IBI325
  Interventions: Drug: IBI363
- IBI363 DL3 (Experimental): IBI363 + Lenvatinib
  Interventions: Drug: IBI363
- IBI363 DL4 (Experimental): IBI363 + Lenvatinib
  Interventions: Drug: IBI363
- IBI363 DL5 (Experimental): Patients with histopathologically confirmed advanced melanoma, who have failed PD-1/PD-L1 treatment and CD73 ≥++ confirmed by IHC.
  Interventions: Drug: IBI363
- IBI363 DL6 (Experimental): Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment and CD73 ≥++ confirmed by IHC.
  Interventions: Drug: IBI363
- IBI363 DL7 (Experimental): Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment, and whose best response during PD-1/PD-L1 treatment was disease stabilization for less than 6 months or disease progression.
  Interventions: Drug: IBI363
- IBI363 DL8 (Experimental): Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment, and whose best response during PD-1/PD-L1 treatment was partial response or complete response lasting more than 6 months.
  Interventions: Drug: IBI363
- IBI363 DL9 (Experimental): Patients with histologically confirmed advanced NSCLC, who have undergone NGS testing confirming the presence of an ALK fusion mutation and have previously failed standard treatment.
  Interventions: Drug: IBI363
- IBI363 DL10 (Experimental): Patients with histological or cytological confirmation of advanced NSCLC who harboring EGFR mutation and failed standard treatment.
  Interventions: Drug: IBI363
- IBI363 DL11 (Experimental): Patients with histological or cytological confirmation of advanced NSCLC and failed standard treatment with rare mutations, including but not limited to ROS1, BRAF V600E, METex14 skipping, HER2, NTRK, and RET fusion.
  Interventions: Drug: IBI363

INTERVENTIONS:
Drug: IBI363 — IBI363 is based on the "3+3" model with a dose of 1 mg/kg Q3W. IBI325, 20 mg/kg Q3W.
  Other Names: IBI325
  Arms: IBI363 DL1
Drug: IBI363 — IBI363 is based on the "3+3" model with a dose of 1.5 mg/kg Q3W. IBI325, 20 mg/kg Q3W.
  Other Names: IBI325
  Arms: IBI363 DL2
Drug: IBI363 — IBI363 is based on the "3+3" model with a dose of 600 μg/kg Q2W. Lenvatinib, 8mg QD.
  Other Names: Lenvatinib
  Arms: IBI363 DL3
Drug: IBI363 — IBI363 is based on the "3+3" model with a dose of 1000 μg/kg Q2W. Lenvatinib, 8mg QD.
  Other Names: Lenvatinib
  Arms: IBI363 DL4
Drug: IBI363 — The recommended dosages for IBI363, IBI325, and Lenvatinib in Phase Ib will be determined based on a comprehensive assessment of safety, efficacy, and other data obtained from the safety introduction portions of both Phase Ia (Part A) and Phase Ib (Part B).
  Arms: IBI363 DL10; IBI363 DL11; IBI363 DL5; IBI363 DL6; IBI363 DL7; IBI363 DL8; IBI363 DL9

SUMMARY:
The study is a prospective multi-cohort clinical study. The study is divided into two phases, Phase Ia and Phase Ib. In Phase Ia, a dose escalation portion was conducted using a 3+3 dose-escalation design, with a preference for enrolling subjects with advanced non-small cell lung cancer and melanoma. Phase Ib represents the cohort expansion phase, comprising seven cohorts.

DETAILED DESCRIPTION:
The study is a prospective multi-cohort clinical study. The study is divided into two phases, Phase Ia and Phase Ib. In Phase Ia, a dose escalation portion was conducted using a 3+3 dose-escalation design, with a preference for enrolling subjects with advanced non-small cell lung cancer and melanoma. Phase Ib represents the cohort expansion phase, comprising seven cohorts. All the research data were collected follow the SAP.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any trial-related procedures
* Age ≥18 years old and ≤75 years old;
* No limit on the gender;
* Phase Ia: Enrollment priority is given to subjects with advanced non-small cell lung cancer and melanoma.
* Phase Ib: This study comprises seven cohorts, including:
* Cohort A: Patients with histopathologically confirmed advanced melanoma, who have failed PD-1/PD-L1 treatment and CD73 ≥++ confirmed by IHC.
* Cohort B: Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment and CD73 ≥++ confirmed by IHC.
* Cohort C: Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment, and whose best response during PD-1/PD-L1 treatment was disease stabilization for less than 6 months or disease progression.
* Cohort D: Patients with histopathologically confirmed advanced NSCLC, who have failed PD-1/PD-L1 treatment, and whose best response during PD-1/PD-L1 treatment was partial response or complete response lasting more than 6 months.
* Cohort E: Patients with histologically confirmed advanced NSCLC, who have undergone NGS testing confirming the presence of an ALK fusion mutation and have previously failed standard treatment.
* Cohort F: Patients with histological or cytological confirmation of advanced NSCLC who harboring EGFR mutation and failed standard treatment.
* Cohort G: Patients with histological or cytological confirmation of advanced NSCLC and failed standard treatment with rare mutations, including but not limited to ROS1, BRAF V600E, METex14 skipping, HER2, NTRK, and RET fusion.
* Tumor assessment according to RECIST v1.1, at least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* 1. Known history of seizures, active central nervous system metastasis, spinal cord compression, carcinomatous meningitis, history of meningeal metastasis, and newly diagnosed brain metastasis or meningeal metastasis.
* a) Subjects who have previously received treatment for central nervous system metastases must meet all of the following criteria to be eligible for this study:
* Completed treatment for central nervous system metastases (e.g., whole-brain radiation therapy, stereotactic radiosurgery, or equivalent treatment) at least 14 days before the first dose of the investigational drug.
* Post-treatment repeat imaging confirmed no evidence of new brain metastases or enlargement of existing brain metastatic lesions (with an interval of ≥4 weeks and using the same imaging technique as the pre-treatment head imaging).
* No requirement for steroid treatment and stable symptoms for at least 14 days before the first dose of the investigational drug.

  b) Subjects who have not previously received treatment for central nervous system metastases must meet all of the following criteria to be eligible for this study:
* No symptoms related to central nervous system metastases.
* Investigator assessment that immediate treatment for central nervous system metastases is not required.
* A maximum of three central nervous system metastatic lesions, with each lesion having a maximum diameter of ≤5 mm.
* 2. Significant cardiovascular and cerebrovascular diseases, including:

  1. Requiring medical intervention due to ventricular arrhythmias or other uncontrolled arrhythmias, such as treatment with anti-arrhythmic drugs.
  2. Severe conduction disturbances (e.g., third-degree atrioventricular block).
  3. HR-corrected QT interval (QTc interval, calculated using the Fridericia method) ≥480 ms.
  4. Uncontrolled hypertension (systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg), a history of hypertensive crisis, or hypertensive encephalopathy.
  5. A history of myocarditis.
  6. Symptomatic congestive heart failure (New York Heart Association functional classes II-IV) or cardiac ultrasound findings indicating left ventricular ejection fraction (LVEF) <50%.
  7. Any arterial thrombosis, embolism, or ischemic event (e.g., myocardial infarction, unstable angina, cerebrovascular accident) within 6 months prior to the first dose of the investigational drug.
  8. History of deep venous thrombosis or any other serious thromboembolic event within the 3 months before enrollment (implantable venous access port or catheter-related thrombosis, or superficial venous thrombosis are not considered "serious" thromboembolic events).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Up to 90 days post last dose
  Number of participants experiencing clinical and laboratory adverse events (AEs)
ORR | 1 year
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, Principal Investigator — Hunan Cancer Hospital; Nong Yang, Principal Investigator — Hunan Cancer Hospital; Xiang Chen, Principal Investigator — Xiangya Hospital of Central South University; Hong Liu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China